CLINICAL TRIAL: NCT06100848
Title: The Impact of Hydrogen Peroxide (H₂O₂) Fumigation on Bacterial Level in Dental Office Environment: A Clinical Trial Investigation
Brief Title: Hydrogen Peroxide Fumigation in Dental Office Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Jacek Matys, Principal Investigator, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WroclawMU5
Record Dates: First submitted 2023-10-12; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Bacterial Infections; Dental Caries; Aerosol Disease
MeSH Terms: conditions — Bacterial Infections; Dental Caries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caries treatment (Active Comparator): The Koch sedimentation method was used to evaluate the aerobic bacterial content in the dental office air. Thirty plates were opened and then sealed 40 minutes after the initiation of caries treatment.
  Interventions: Diagnostic Test: Microbiological analysis after Caries treatment
- Caries treatment and fumigation (Active Comparator): The Koch sedimentation method was employed to evaluate the aerobic bacterial content in the dental office air. Thirty plates were opened and subsequently sealed 60 minutes after the commencement of caries treatment. Fumigation was conducted for 20 minutes.
  Interventions: Diagnostic Test: Microbiological analysis after Caries treatment and fumigation

INTERVENTIONS:
Diagnostic Test: Microbiological analysis after Caries treatment — Microbiological analysis was conducted for 30 patients using 30 microbiological plates. These plates were opened simultaneously with the start of the treatment and closed 40 minutes later.
  Arms: Caries treatment
Diagnostic Test: Microbiological analysis after Caries treatment and fumigation — Microbiological analysis was conducted for 30 patients using 30 microbiological plates. These plates were opened simultaneously with the start of the treatment and closed 60 minutes later (when fumigation was finished)
  Arms: Caries treatment and fumigation

SUMMARY:
The study's null hypothesis posits no significant difference in bacterial levels in the dental office environment before and after implementing hydrogen peroxide (H₂O₂) fumigation. The study comprised 30 participants, 18 females and 12 males, all diagnosed with moderate caries decay (ICDAS 3 and 4) in their mandibular molars, averaging 42.2 ± 8.3 years in age. Sample size calculations for 30 microbiological plates in each group utilized G*Power software (Kiel University, Germany), factoring in prior research, with a significance level of 0.05, effect size (d) of 0.72, 95% confidence interval, and 85% power. Aerobic bacterial content in the dental office air was assessed using the Koch sedimentation method. The study employed 60 Petri dishes with Columbia Agar and 5% Sheep Blood. During caries treatment, thirty plates were opened and sealed 40 minutes later, while another set of thirty plates was opened and closed 60 minutes post-fumigation. Measurements were taken 1 meter above the ground and 2 meters from the patient's mouth. After 48 hours of incubation at 37°C, microbiological contamination was calculated as CFUs (colony-forming units) in one cubic meter using the formula: L = a × 1000 / (πr² × k). Fumigation involved a 20-minute treatment with 6% hydrogen peroxide biosanitizer (Saniswiss, Switzerland) via a compressed air device (Fumi-Jet, Kormed, Poland). The process included 3 minutes of fumigation and a 17-minute waiting period for the chemotoxic effect, with 45 ml of 6% hydrogen peroxide sprayed in a 20 m² room.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with moderate caries decay based on the International Caries Detection and Assessment System (ICDAS 3 and 4) in their mandibular molar teeth
* received hygienist treatment two weeks before the study initiation

Exclusion Criteria:

* use anti-inflammatory medications
* non-smokers
* had systemic illnesses
* with uncompensated diabetes
* with halitosis symptoms
* with gastric diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Number of bacteria after caries treatment | After 48 hours of incubation
  At the onset of caries treatment, thirty plates (n=30) will be opened and will be sealed 40 minutes later.
  After 48 hours of incubation at 37°C, the degree of microbiological contamination will be determined, calculated as the total number of CFUs (colony-forming units) in one cubic meter of air using the formula: L = a × 1000 / (πr² × k). In the formula, L represents the microbial contamination level in [cfu/m3], 'a' signifies the quantity of bacterial colonies cultivated on the plate, 'r' denotes the Petri dish radius [cm], and 'k' stands for the plate exposure time factor, with k = t × 1/5, where 't' represents the exposure time in minutes.
Number of bacteria after caries treatment and fumigation | After 48 hours of incubation
  Another set of thirty plates (n=30) will be opened immediately before caries treatment and closed 60 minutes later following the completion of fumigation. After 48 hours of incubation at 37°C, the degree of microbiological contamination will be determined, calculated as the total number of CFUs (colony-forming units) in one cubic meter of air using the formula: L = a × 1000 / (πr² × k). In the formula, L represents the microbial contamination level in [cfu/m3], 'a' signifies the quantity of bacterial colonies cultivated on the plate, 'r' denotes the Petri dish radius [cm], and 'k' stands for the plate exposure time factor, with k = t × 1/5, where 't' represents the exposure time in minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Oral Surgery Department, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No